CLINICAL TRIAL: NCT04618861
Title: Surfactant Protein D Levels in Covid-19 Infection: Case-Control Study
Status: Completed | Type: Observational
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Ramazan Sbirli, Dr., Kafkas University
Other Study IDs: Clinical-1
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Pneumonia; Surfactant Protein Deficiency
Keywords: Serum surfactant protein D; SARS-CoV-2 infection; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Only serum specimens will be analyze for meassuring the level of the serum surfactant protein D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control Group: This cohort involved the volunteers who had no known acute, subacute or chronic disease history, who did not suffer from any infection in the last fortnight, who were not on a particular medication, who presented to the ED with reasons other than infectious complaints, and who gave their written consent to participate in the study.
  The exclusion criteria consisted of diagnosis of kidney and liver failure, acute pulmonary embolism, chronic inflammatory disease history (rheumatological disease, autoimmune disease), pregnancy, presence of any cancer diagnosis, chronic obstructive pulmonary disease, asthma disease, and history of cerebrovascular disease. In addition, the patients whose CT imagings were compatible with Covid-19 pneumonia but whose PCR tests were negative were also excluded from the study.
- CT (+), PCR (-) Covid-19 Suspected Pneumonia Group: This group consisted of patients who applied to the emergency department with symptoms of Covid-19, whose thorax CT according to RSNAEC criteria showed typical Covid-19 pneumonia findings, but whose RT-PCR test was negative in the swab sample taken in the emergency room.
  The exclusion criteria consisted of diagnosis of kidney and liver failure, acute pulmonary embolism, chronic inflammatory disease history (rheumatological disease, autoimmune disease), pregnancy, presence of any cancer diagnosis, chronic obstructive pulmonary disease, asthma disease, and history of cerebrovascular disease. In addition, the patients whose CT imagings were compatible with Covid-19 pneumonia but whose PCR tests were negative were also excluded from the study.
- CT (+), Covid-19 Pneumonia Group: This cohort consisted of the patients (a) who applied to the emergency department with SARS-CoV-2 symptoms and was diagnosed with SARS-CoV-2 infection according to WHO guideline (13) (b) whose CT imagings were compatible with SARS-CoV-2 pneumonia in accordance with the Radiological Society of North America Expert Consensus (RSNAEC) criteria (14), (c) whose nasopharyngeal swab samples taken in the ED were positive for RT-PCR, and (d) who gave their informed consent to participate in the study.
  The exclusion criteria consisted of diagnosis of kidney and liver failure, acute pulmonary embolism, chronic inflammatory disease history (rheumatological disease, autoimmune disease), pregnancy, presence of any cancer diagnosis, chronic obstructive pulmonary disease, asthma disease, and history of cerebrovascular disease. In addition, the patients whose CT imagings were compatible with Covid-19 pneumonia but whose PCR tests were negative were also excluded from the study.
- CT (-), PCR (+) Covid-19 infection group: This cohort included the patients (a) who presented to the Covid-19 outpatient polyclinic of the ED with pneumonia symptoms, (b) whose CT imaging's were compatible with Covid-19 pneumonia in accordance with the RSNAEC criteria and whose PCR tests were positive, (c) whose SARS-CoV-2 PCR tests were positive as a result of contact tracing, and (d) who presented to the ED for further examination.
  The exclusion criteria consisted of diagnosis of kidney and liver failure, acute pulmonary embolism, chronic inflammatory disease history (rheumatological disease, autoimmune disease), pregnancy, presence of any cancer diagnosis, chronic obstructive pulmonary disease, asthma disease, and history of cerebrovascular disease. In addition, the patients whose CT imagings were compatible with Covid-19 pneumonia but whose PCR tests were negative were also excluded from the study.

SUMMARY:
This study aims to provide some insight into the variation of SD-D protein levels in patients with Covid-19 (-) pneumonia, Covid-19 (+) pneumonia, and CT negative Covid-19 infection in comparison to the normal population through a larger number of cases. Objective of the study is to determine the serum surfactant protein D (SP-D) levels in Covid-19 pneumonia infection.

DETAILED DESCRIPTION:
This study aims to provide some insight into the variation of SD-D protein levels in patients with Covid-19 (-) pneumonia, Covid-19 (+) pneumonia, and CT negative Covid-19 infection in comparison to the normal population through a larger number of cases. Subjects will assessed in accordance with the inclusion and exclusion criteria, they were divided into four groups as the CT (-), PCR (+) SARS-CoV-2 infection group, SARS-CoV-2 (+) Pneumonia Group, CT (+), PCR (-) Suspected Pneumonia Group and Healthy group (Control Group). Demographic data, medical history, vital findings (fever, blood pressure, sPO2), laboratory findings (complete blood count; C-reactive protein (CRP), D-dimer, Ferritin and hsTnT parameters) and radiological findings, time to onset of symptoms, Comorbid diseases, hospitalization location of the patients (service or ICU), clinical scores, CT severity scores will determine. SP-D level will analyze by the Enzyme-Linked Immunosorbent Assay (ELISA) method.

ELIGIBILITY:
For patients;

Inclusion Criteria:

* who presented to the Covid-19 outpatient polyclinic of the ED with pneumonia symptoms,
* whose CT imaging's were compatible with Covid-19 pneumonia in accordance with the RSNAEC criteria and whose PCR tests were positive,
* whose SARS-CoV-2 PCR tests were positive as a result of contact tracing,
* who presented to the ED for further examination.
* who gave their written consent to participate in the study.
* Giving written consent to participate in the study.

Exclusion Criteria:

* diagnosis of kidney or liver failure
* acute pulmonary embolism
* chronic inflammatory disease history (rheumatological disease, autoimmune disease),
* pregnancy
* presence of any cancer diagnosis
* chronic obstructive pulmonary disease
* asthma disease,
* history of cerebrovascular disease.
* the patients whose CT imagings were compatible with Covid-19 pneumonia but whose PCR tests were negative were also excluded from the study.

For control group Inclusion Criteria

* no known acute, subacute or chronic disease history
* not suffer from any infection in the last fortnight,
* not to be on a particular medication,
* Presenting to the ED with reasons other than infectious complaints
* Giving written consent to participate in the study.

Exclusion Criteria:

* diagnosis of kidney or liver failure
* acute pulmonary embolism
* chronic inflammatory disease history (rheumatological disease, autoimmune disease),
* pregnancy
* presence of any cancer diagnosis
* chronic obstructive pulmonary disease
* asthma disease,
* history of cerebrovascular disease.

Min Age: 18 Years
Age Groups: Adult, Older Adult
Study Population: After the required information concerning the study was provided both to the patient group and to the healthy control group, the written consent forms were obtained from all the subjects who agreed to participate in the study.
  Once these subjects were assessed in accordance with the inclusion and exclusion criteria. Patients who were diagnosed with Covid-19 infection according to WHO guideline as a result of clinical evaluation in the emergency department and whose diagnosis was confirmed by RT-PCR were included in the study.
  The healthy volunteers with no known chronic or acute disease or drug use as well as no recent history of infection were included study as the control group. Once these subjects were assessed in accordance with the inclusion and exclusion criteria, they were divided into four groups as the CT (-), PCR (+) SARS-CoV-2 infection group, Covid-19 (+) Pneumonia Group, CT (+), PCR (-) Suspected Pneumonia Group and Healthy group (Control Group).
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Meassuring the serum surfactant protein D levels in patient who have Covid-19 infection or pneumonia. | 2 months
  First primary outcome is determining the serum surfactant protein D level changes in patient who have Covid-19 infection or pneumonia aganist healty controls.
Analyzing the correlations between serum surfactant protein D levels and demographic,laboratory, clinical and radiological datas. | 2 months
  Determining the correlation between between serum surfactant protein D levels and demographic datas (age,gender), medical history, vital findings (fever, blood pressure, sPO2), laboratory findings (complete blood count; C-reactive protein (CRP), D-dimer, Ferritin and hsTnT parameters) and radiological findings, time to onset of symptoms, Comorbid diseases, hospitalization location of the patients (service or ICU), clinical scores (PSI and CURB65 scores), CT severity scores .

CONTACTS AND LOCATIONS:
Locations (1):
- Aylin Koseler, Denizli, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing the patient datas.